CLINICAL TRIAL: NCT01458223
Title: The Effect of Prolonged Postoperative Antibiotics Administration on Rate of Infection in Patients Undergoing Posterior Spine Surgery Requiring a Hemovac Drain
Acronym: PARISS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The London Spine Centre (Other)
Responsible Party: Principal Investigator, Dr. Christopher Bailey, Principal Investigator, The London Spine Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17846
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Infection
Keywords: spine surgery; postoperative infection; postoperative antibiotics
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): 24 hours post-operative antibiotics
  Interventions: Drug: Antibiotic
- experimental (Experimental): 72 hours of post-operative antibiotics
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Drug: Antibiotic — Ancef or Vancomycin
  Arms: Control
Drug: Antibiotic — Ancef or Vancomycin
  Arms: experimental

SUMMARY:
Post-operative antibiotics for infection prophylaxis are routinely given to most surgical patients, and for orthopaedic surgery patients, the standard of care is treatment for 24 hours following any elective procedure (1). The most concerning risk for insufficient antibiotic coverage in the post-operative period is the development of a complicated infection requiring irrigation and debridement or revision surgery. Moreover, recovery from surgery is usually delayed in patients that have postoperative wound infections leading to increased resource utilization and increased economic cost for the health care system. It is clear that prophylactic antibiotic therapy is necessary in the immediate post-operative period, but the length required continues to be debated.

Orthopaedic patients undergoing elective spine surgeries often require the placement of a hemovac drain which applies gentle suction to remove excess fluid/blood and to promote healing. Wound drains, however, may also increase the risk of post-operative infection because they expose the "clean" interior aspect of the wound to the "dirty" exterior area around the wound. Given this additional focus of infection, it is unknown whether prolonged antibiotic therapy post-operatively is needed to decrease the rate of infection in this population (2,3). There is sparse literature evaluating the effectiveness of prolonged antibiotic therapy in decreasing complicated post-operative infection requiring irrigation and debridement in this population (1,4). To our knowledge, there are no recent studies comparing prophylactic antibiotics for 24 hours only post-operatively versus 24 hours after removal of the drain. In fact, a recent evidence-based review of the literature by the North American Spine Society highlighted the need for research in this area (5).

The proposed study will compare two patient populations who will receive various lengths of post-operative antibiotics. One will receive only 24 hours worth, and the other will receive antibiotics for 72 hours after surgery and the rate of complicated infection compared between the two.

The absence of a demonstrable difference suggests that antibiotic prophylaxis for only 24 hours immediately post-operatively is sufficient for all elective spine patients undergoing posterior spine procedures requiring the placement of a hemovac drain.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 and older
* Require spine surgery for posterior lumbar decompressions, posterior thoracic decompressions, posterior cervical decompressions, posterior lumbar fusions, posterior thoracic fusions, posterior cervical fusions
* English speaking and able to understand and provide informed consent

Exclusion Criteria:

* Known hypersensitivity to antibiotics
* Severe renal function impairments
* Antibiotic therapy for concomitant infection at the time of surgery
* Spine patients not requiring the insertion of a hemovac drain
* Pregnant
* Concomitant steroid therapy
* Permanent residence more than a 5 hour driving distance away from Hospital

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Infection Rate | one year
  complicated wound infection requiring surgical irrigation and debridement

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital, London Health Sciences Centre, London, Ontario, Canada